CLINICAL TRIAL: NCT05889858
Title: Medical Follow-up of Medical Secretaries of General Practitioners
Acronym: Suivi-secret
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_002_Suivi-Secret
Record Dates: First submitted 2023-05-11; First posted 2023-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Medical Follow-up of Medical Secretaries
Keywords: medical secretaries; general practitioners; medical follow-up
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "medical secretaries of general practitioners" group: Men and women working as a secretary for a general practitioner, face-to-face in the medical practice.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
General practitioners are very often confronted with requests for care from their relatives (family, friends, etc.). In the United States, the recommendations advise general practitioners against taking care of their loved ones on several grounds: lack of professional objectivity, lack of information due to modesty, risk of loss of patient autonomy. Some countries even prohibit general practitioners from prescribing to a loved one except in an emergency.

In France, there is no current recommendation on the care of relatives. Half of French general practitioners have a physical secretary and are therefore potentially confronted with requests for care from their medical secretary.

DETAILED DESCRIPTION:
The aim of the study is to describe the medical follow-up of medical secretaries of general practitioners

ELIGIBILITY:
Inclusion Criteria:

* medical secretaries of general practitioners
* work in face-to-face in the medical practice
* agreed to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: medical secretaries of general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
type of attending physician | Day 1
  type of attending physician will be either the general practitioner employing the medical secretary or an another physician (an another general practitioner or a specialist)

CONTACTS AND LOCATIONS:
Overall Officials: Hurtaud Aline, Dr, Principal Investigator — Université Reims Champagne-Ardenne
Locations (1):
- Université de Reims Champagne Ardenne, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided